CLINICAL TRIAL: NCT02002533
Title: Feasibility, Acceptability and Mechanisms of Brief Behavioral Therapy (BBT) for Sleep Problems During Chemotherapy: A Phase II Randomized Controlled Trial
Brief Title: Brief Behavioral Therapy in Improving Sleep Disorders in Patients With Stage I-III Breast Cancer Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gary Morrow (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Stanford University (Other)
Responsible Party: Sponsor-Investigator, Gary Morrow, Director, University of Rochester NCORP Research Base
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: URCC12048; NCI-2013-01170 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); URCC12048 (Other: University of Rochester); URCC-12048 (Other: DCP); URCC12048 (Other: CTEP); UG1CA189961 (NIH); U10CA037420 (NIH)
Record Dates: First submitted 2013-11-30; First posted 2013-12-06 (Estimated); Results first posted 2017-12-02 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Sleep Disorder; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Sleep Wake Disorders; Breast Neoplasms | interventions — Behavior Therapy; Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (BBT intervention) (Experimental): Patients undergo BBT intervention, comprising insomnia education, stimulus control, discouragement of napping and encouragement of exercise, and sleep compression over two 60 minute face-to-face sessions in weeks 1 and 3 or 4, and four 15 minute telephone sessions in weeks 2, 3, 5, and 6 or 2, 4, 5, and 6.
  Interventions: Behavioral: Brief Behavioral Therapy; Behavioral: Telephone-Based Intervention
- Arm II (control) (Active Comparator): Patients undergo HEAL comprising nutritional education and suggestions for symptom management over two 60 minute face-to-face sessions in weeks 1 and 3 or 4, and four 15 minute telephone sessions in weeks 2, 3, 5, and 6 or 2, 4, 5, and 6.
  Interventions: Other: Educational Intervention; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Behavioral: Brief Behavioral Therapy — Undergo BBT intervention
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions
  Arms: Arm I (BBT intervention)
Behavioral: Telephone-Based Intervention — Undergo BBT intervention
  Arms: Arm I (BBT intervention)
Other: Educational Intervention — Undergo HEAL
  Other Names: Education for Intervention; Intervention, Educational
  Arms: Arm II (control)
Behavioral: Telephone-Based Intervention — Undergo HEAL
  Arms: Arm II (control)

SUMMARY:
This randomized phase II trial studies how well brief behavioral therapy works in improving sleep disorders in patients with stage I-III breast cancer undergoing chemotherapy. Sleep disorder counseling may reduce fatigue and insomnia as well as improve the well-being and quality of life in patients with breast cancer who are undergoing chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine recruitment rates to the proposed randomized controlled trial (RCT).

II. Determine the rate of intervention adherence. III. Determine the feasibility of training National Cancer Institute (NCI) Community Oncology Research Program (NCORP) clinical research staff to successfully deliver the Brief Behavioral Therapy (BBT) intervention.

SECONDARY OBJECTIVES:

I. Obtain preliminary estimates for the effect of the intervention (compared with control) on insomnia as measured by the Insomnia Severity Index (ISI).

II. Obtain preliminary estimates for the effect of the intervention (compared with control) on sleep quality as measured by the Pittsburgh Sleep Quality Index (PSQI).

III. Obtain preliminary estimates for the effect of the intervention (compared with control) on circadian rhythm as measured by the two-oscillator cosinor parameter estimates based on actigraphy data.

IV. Obtain preliminary estimates for the effect of the intervention (compared with control) on heart rate variability (HRV) as measured by the Firstbeat® ambulatory heart-rate monitor (i.e., 1. respiratory sinus arrhythmia-RSA, 2. standard deviation of all normal R-wave to R-wave intervals--SDNN, 3. root mean square of successive differences between adjacent normal R-wave to R-wave intervals--RMSSD, 4. The ratio of low frequency total spectrum power of all NN intervals between .04 to .15 Hertz to high frequency total spectrum power of all NN intervals between .15 to .40 Hertz--LF/HF ratio, and 5. natural log of low frequency total spectrum power of all NN intervals between 0.04 to 0.15Hz.).

TERTIARY OBJECTIVES:

I. Obtain preliminary estimates for the effect of the intervention (compared with control) on quality of life as measured by the Functional Assessment of Chronic Illness Therapy (FACIT) total score and subscales.

II. Obtain preliminary estimates for the effect of the intervention (compared with control) on general mood as measured by the Profile of Mood States (POMS) total score and subscales.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo BBT intervention, comprising insomnia education, stimulus control, discouragement of napping and encouragement of exercise, and sleep compression over two 60 minute face-to-face sessions in weeks 1 and 3 or 4, and four 15 minute telephone sessions in weeks 2, 3, 5, and 6 or 2, 4, 5, and 6.

ARM II: Patients undergo Healthy Eating Education (HEAL) comprising nutritional education and suggestions for symptom management over two 60 minute face-to-face sessions in weeks 1 and 2 or 3, and four 15 minute telephone sessions in weeks 2, 3, 5, and 6 or 2, 4, 5, and 6.

After completion of study, patients are followed up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed breast cancer (stage I, II, III)
* Be receiving chemotherapy in either weekly, 2-week or 3-week cycles and have at least 6 weeks of chemotherapy treatment remaining; patients are eligible any time before chemotherapy cycle 3 if on a 2- or 3-week cycle, or cycle 4 if on a 1-week cycle; (Note: use of biologics [e.g., Herceptin (trastuzumab)] is permitted)

  * For patients on a weekly regimen, there should be at least 3 dosages of chemotherapy remaining
  * For patients on either a 2 week or 3 week cycle, there should be at least 2 dosages of chemotherapy remaining
  * Patients will not be dropped from the study if their chemotherapy is discontinued after they are enrolled
* Report sleep disturbance of 8 (sum total of all 7 items) or greater on the Insomnia Severity Index

  * (Note: this measure will be repeated again at baseline assessment)
* Report sleep problems that began or got worse with the diagnosis of cancer or with chemotherapy; (did your sleep problems begin or get worse with the diagnosis of cancer or with chemotherapy?)
* Be able to speak and read English
* Patients can take sleep aids (e.g., hypnotics and sedatives) for insomnia if they use sleep aids as needed; patients taking sleep aids every night are excluded; use of melatonin every night is permitted and these patients are not excluded
* Be able and willing to wear an Actiwatch for the entire 24 hours of each day they are scheduled to wear it

Exclusion Criteria:

* Have diagnosis of breast cancer stage IV
* Have sleep problems that began before diagnosis and have not changed since diagnosis
* Self-report or have a medical record of an unstable comorbid medical or psychiatric condition that would make it unsafe or impossible to adhere to the study protocol
* Have a clinical diagnosis of sleep apnea or restless leg syndrome
* Be unable or unwilling to discontinue anxiolytic medication within 4 hours of intervention sessions
* Take medication for sleep (e.g., hypnotics and sedatives) every night; melatonin is permitted
* Patients who are shift workers are excluded; shift worker is defined as someone who has irregular work and sleep hours (such as working a non-traditional schedule: e.g., 4pm-midnight or 10pm-6am; a rotating schedule e.g., alternating between day and night shifts, or starting work between 4am and 7am)
* Have an implanted device for heart failure (e.g., pacemaker, defibrillator, left ventricular assist device, etc.)

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-02-03 (Actual); Primary Completion 2016-12-16 (Actual); Study Completion 2016-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oxana Palesh, Principal Investigator — University of Rochester NCORP Research Base
Locations (6):
- United States (6):
  - Stanford University Medical Center, Stanford, California
  - Heartland NCORP, Decatur, Illinois
  - Wichita NCORP, Wichita, Kansas
  - Metro-Minnesota NCORP, Minneapolis, Minnesota
  - University of Rochester, Rochester, New York
  - Southeast Clinical Oncology Research Program, Winston-Salem, North Carolina

REFERENCES:
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (BBT Intervention) | Arm II (Control)
Started | 34 | 37
Completed | 28 | 19
Not Completed | 6 | 18
Not completed — Withdrawal by Subject | 6 | 13
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 0 | 3
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (BBT Intervention) | Arm II (Control) | Total
Number analyzed (Participants) | 34 | 37 | 71
Age, Continuous [Mean (Full Range); unit: years] | 50.9 [33 to 67] | 53.9 [29 to 73] | 52.5 [29 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 37 | 71
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 34 | 37 | 71
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 33 | 35 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 37 | 71

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eligible Patients Consented
Description: Will be evaluated by calculating the specific percentage (with 95% confidence interval) of the total number of participants approached that then consented and enrolled in the study.
Time Frame: baseline
Population: 92 people were approached to enroll in the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All Participants: All people that were enrolled in the study regardless of intervention assigned.
Arm/Group | All Participants
Number analyzed (Participants) | 92
percentage of participants | 77.17 [67.61 to 84.55]
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p > 0.9999, exact binomial test; The percentage is greater than or equal to 40%

2. Primary Outcome: Percentage of Consented Participants Who Complete the Study, Defined as Completion of at Least 5 BBT
Description: Will be evaluated by calculating the specific percentage (with 95% confidence interval) and performing an exact binomial test with the null hypothesis being greater than or equal to 75%.
Time Frame: Up to 1 month
Population: Data on HEAL subjects was not collected since the main focus was BBT, therefore only rate of adherence is shown for BBT group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (BBT Intervention) | Arm II (Control)
Number analyzed (Participants) | 34 | 0
percentage of participants | 73.5 [55.3 to 86.5] |
Statistical Analysis 1: Comparison: Arm I (BBT Intervention); Test type: Superiority; p = 0.7350, exact binomial test

3. Primary Outcome: Percentage of Key Components of BBT Delivered by NCI Community Oncology Research Program (NCORP) Staff, Assessed by Checklist and Auditing of Audio-recordings
Description: Each NCORP staff person completed a study checklist in which they designated which concepts they discussed with the patient at each session. Concepts included how sleep problems develped, how to control stimulus, and sleeping environment. The overall mean percent delivery was measured using a random effects model (residual maximum likelihood [REML] estimation), where the intercept represents the mean delivery and three independent random effects are included. Because of the small sample size, testing will use the Kenward-Roger procedure.
Time Frame: Up to 1 month
Population: This assessment was only performed for the BBT arm.
Measure: Mean (Standard Error); unit: percentage of components delivered
Arm/Group | Arm I (BBT Intervention) | Arm II (Control)
Number analyzed (Participants) | 34 | 0
percentage of components delivered | 0.8075 (0.08450) |
Statistical Analysis 1: Comparison: Arm I (BBT Intervention); Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.8075, Standard Error of Mean 0.08450

4. Secondary Outcome: Change in Insomnia as Measured by the Insomnia Severity Index (ISI)
Description: The ISI has seven questions. The seven answers are added up to get a total score.
  Total score categories:
  0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe) The difference between arms will be assessed using analysis of covariance (ANCOVA). The response will be the post-intervention outcome. Arm will be the factor, and baseline will be the covariate. Appropriate contrasts will be used to estimate the difference between arms in change from baseline. Initially, the arm*baseline interaction will be assessed with an F test. If this interaction is insignificant at the 0.05 level, it will be dropped from the final model. If the interaction is significant, then mean change from baseline at various levels of baseline will be reported.
Time Frame: Baseline to up to 1 month
Population: Based on subjects that completed study through post-intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (BBT Intervention) | Arm II (Control)
Number analyzed (Participants) | 28 | 19
units on a scale | -6.259 (5.134) | -2.450 (6.700)
Statistical Analysis 1: Comparison: Arm I (BBT Intervention) vs Arm II (Control); Test type: Superiority; p = 0.1808, ANCOVA; Mean Difference (Final Values) = -1.64, Standard Error of Mean 1.21 — The estimated value is BBT minus HEAL

5. Secondary Outcome: Change in Sleep Quality as Measured by the Pittsburgh Sleep Quality Index (PSQI)
Description: Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality. The difference between arms will be assessed using ANCOVA. The response will be the post-intervention outcome. Arm will be the factor, and baseline will be the covariate. Appropriate contrasts will be used to estimate the difference between arms in change from baseline. Initially, the arm*baseline interaction will be assessed with an F test. If this interaction is insignificant at the 0.05 level, it will be dropped from the final model. If the interaction is significant, then mean change from baseline at various levels of baseline will be reported.
Time Frame: Baseline to up to 1 month
Population: Based on subjects that completed study through post-intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (BBT Intervention) | Arm II (Control)
Number analyzed (Participants) | 28 | 19
units on a scale | -4.000 (3.590) | -2.750 (4.089)
Statistical Analysis 1: Comparison: Arm I (BBT Intervention) vs Arm II (Control); Test type: Superiority; p = 0.14, ANCOVA; Mean Difference (Final Values) = -1.08, Standard Error of Mean 0.73 — Estimated value is BBT minus HEAL

6. Secondary Outcome: Change in Mean Circadian Rhythm Mesor
Description: Activity levels were measured using an actigraphy device worn as a watch. The data was collected by the device for a 24 hour period. A model consisting of two cosine functions, one with a period of 12 hours, and the other with a period of 24 hours is fit to log activity counts as the dependent variable, and hour (0 to 24) as the independent variable. The mesor is the average activity over a 24 hour period.
Time Frame: Baseline to up to 1 month
Population: Based on subjects that completed study through post-intervention.
Measure: Mean (Standard Deviation); unit: log activity counts
Arm/Group | Arm I (BBT Intervention) | Arm II (Control)
Number analyzed (Participants) | 28 | 19
log activity counts | 0.008 (0.153) | -0.046 (0.156)
Statistical Analysis 1: Comparison: Arm I (BBT Intervention) vs Arm II (Control); Test type: Superiority; p = 0.005, ANCOVA; For baseline of 0.7; Mean Difference (Final Values) = 0.404, Standard Error of Mean 0.137
Statistical Analysis 2: Comparison: Arm I (BBT Intervention) vs Arm II (Control); Test type: Superiority; p = 0.092, ANCOVA — At baseline 1.3; Mean Difference (Final Values) = 0.077, Standard Error of Mean 0.045
Statistical Analysis 3: Comparison: Arm I (BBT Intervention) vs Arm II (Control); Test type: Superiority; p = 0.556, ANCOVA — At baseline of 1.5; Mean Difference (Final Values) = -0.032, Standard Error of Mean 0.053
Statistical Analysis 4: Comparison: Arm I (BBT Intervention) vs Arm II (Control); Test type: Superiority; p = 0.007, ANCOVA — Grouped by baseline interaction; Mean Difference (Final Values) = -6.24, Standard Error of Mean 0.221 — The estimated value is grouped by baseline interaction parameter

7. Secondary Outcome: Change in Circadian Rhythm Amplitude Over 24 Hours
Description: Activity levels were measured using an actigraphy device worn as a watch. The data was collected by the device for a 24 hour period. A model consisting of two cosine functions, one with a period of 12 hours, and the other with a period of 24 hours is fit to log activity counts as the dependent variable, and hour (0 to 24) as the independent variable. The ampliitude is the peak activity level over a 24 hour period.
Time Frame: baseline to up to 1 month
Population: Based on subjects that completed study through post-intervention.
Measure: Mean (Standard Deviation); unit: log10 (counts/minute)
Arm/Group | Arm I (BBT Intervention) | Arm II (Control)
Number analyzed (Participants) | 28 | 19
log10 (counts/minute) | 0.061 (0.185) | -0.164 (0.194)
Statistical Analysis 1: Comparison: Arm I (BBT Intervention) vs Arm II (Control); Test type: Superiority; p = 0.000, ANCOVA

8. Secondary Outcome: Change in Circadian Rhythm Amplitude Over 12 Hours
Description: Activity levels were measured using an actigraphy device worn as a watch. The data was collected by the device for a 24 hour period. A model consisting of two cosine functions, one with a period of 12 hours, and the other with a period of 24 hours is fit to log activity counts as the dependent variable, and hour (0 to 24) as the independent variable. The amplitude is the highest activity level over a 12 hour period.
Time Frame: baseline to up to 1 month
Population: Based on subjects that completed study through post-intervention.
Measure: Mean (Standard Deviation); unit: log10 (counts/minute)
Arm/Group | Arm I (BBT Intervention) | Arm II (Control)
Number analyzed (Participants) | 28 | 19
log10 (counts/minute) | 0.063 (0.164) | 0.127 (0.236)
Statistical Analysis 1: Comparison: Arm I (BBT Intervention) vs Arm II (Control); Test type: Superiority; p = 0.295, ANCOVA

9. Secondary Outcome: Change in Mean Circadian Rhythm Acrophase Over 24 Hours
Description: Activity levels were measured using an actigraphy device worn as a watch. The data was collected by the device for a 24 hour period. A model consisting of two cosine functions, one with a period of 12 hours, and the other with a period of 24 hours is fit to log activity counts as the dependent variable, and hour (0 to 24) as the independent variable. The acrophase is the time where peak activity occurs over a 24 hour period. The larger the acrophase the later in the day is the peak activity.
Time Frame: baseline to up to 1 month
Population: Based on subjects that completed study through post-intervention.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Arm I (BBT Intervention) | Arm II (Control)
Number analyzed (Participants) | 28 | 19
hours | 0.409 (3.698) | -0.912 (2.855)
Statistical Analysis 1: Comparison: Arm I (BBT Intervention) vs Arm II (Control); Test type: Superiority; p = 0.573, ANCOVA

10. Secondary Outcome: Change in Mean Circadian Rhythm Acrophase Over 12 Hours
Description: Activity levels were measured using an actigraphy device worn as a watch. The data was collected by the device for a 24 hour period. A model consisting of two cosine functions, one with a period of 12 hours, and the other with a period of 24 hours is fit to log activity counts as the dependent variable, and hour (0 to 24) as the independent variable. The acrophase is the time where peak activity occurs over a 12 hour period. The larger the acrophase the later in the day is the peak activity.
Time Frame: baseline to up to 1 month
Population: Based on subjects that completed study through post-intervention.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Arm I (BBT Intervention) | Arm II (Control)
Number analyzed (Participants) | 28 | 19
hours | 0.529 (2.519) | 1.516 (4.833)
Statistical Analysis 1: Comparison: Arm I (BBT Intervention) vs Arm II (Control); Test type: Superiority; p = 0.015, ANCOVA; Mean Difference (Final Values) = -6.502, Standard Error of Mean 2.558 — Group difference (BBT - HEAL) in mean post-pre change
Statistical Analysis 2: Comparison: Arm I (BBT Intervention) vs Arm II (Control); Test type: Superiority; p = 0.094, ANCOVA; Mean Difference (Final Values) = -1.723, Standard Error of Mean 1.007 — Group difference (BBT - HEAL) in mean post-pre change
Statistical Analysis 3: Comparison: Arm I (BBT Intervention) vs Arm II (Control); Test type: Superiority; p = 0.114, ANCOVA; Mean Difference (Final Values) = 3.750, Standard Error of Mean 2.326 — Group difference (BBT - HEAL) in mean post-pre change
Statistical Analysis 4: Comparison: Arm I (BBT Intervention) vs Arm II (Control); Test type: Superiority; p = 0.027, ANCOVA; Mean Difference (Final Values) = 0.911, Standard Error of Mean 0.400 — This is an arm by baseline interaction parameter

ADVERSE EVENTS:
Arm/Group | Arm I (BBT Intervention) | Arm II (Control)
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/37
Other Adverse Events (participants affected / at risk) | 0/34 | 3/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (BBT Intervention) (N=34) | Arm II (Control) (N=37)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
mucositis stomastitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
hypotension (Vascular disorders) | 0 (0) | 1 (1)
hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes